CLINICAL TRIAL: NCT01447849
Title: The Impact of Lubiprostone on Mucus Secretion in Asymptomatic Volunteers and Patients With Chronic Constipation
Brief Title: Lubiprostone and Mucus Secretion in Patients With Chronic Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Jerzy Sarosiek, Professor of Medicine, Associate Chairman for Research, Internal Medicine Department, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MSA-LUB-125; MSA-NC-LUB-125 (Other Grant/Funding Number: Takeda Pharmaceuticals); NCT00595036 (obsolete NCT alias)
Record Dates: First submitted 2011-09-14; First posted 2011-10-06 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2015-11

CONDITIONS: Constipation
Keywords: Chronic Constipation
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone 24 mcg Twice a day (Active Comparator): Both controls and patients with chronic constipation will receive 1 week of therapy with lubiprostone and one week of placebo.
  Interventions: Drug: lubiprostone
- Placebo (Placebo Comparator): Both controls and patients with chronic constipation will receive placebo pills twice daily for one week in cross over design
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lubiprostone — 24mcg twice a day (BID) 1 week
  Other Names: Amitiza
  Arms: Lubiprostone 24 mcg Twice a day
Drug: placebo — Placebo pills twice a day for one week.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that the symptoms of chronic constipation in some patients are developed due to diminished production and secretion of the alimentary tract mucus resulting in poor lubrication.

Therefore, the investigators assume that administration of lubiprostone may restore this lubrication impairment by stimulation of mucus production and secretion within the gastrointestinal tract.

DETAILED DESCRIPTION:
Specific Aim 1. To test the effect of Lubiprostone, 24 mcg twice a day (BID) for 1 week, on gastric mucus production in 20 asymptomatic volunteers and 20 patients with chronic constipation in basal conditions (primary outcome).

Specific Aim 2. To explore the effect of Lubiprostone, 24 mcg twice a day (BID) for 1 week, on gastric mucus production in 20 asymptomatic volunteers and 20 patients with chronic constipation during stimulation of gastric secretion with pentagastrin, mimicking the meal-stimulated conditions (primary outcome).

Specific Aim 3. To address the influence of Lubiprostone, 24 mcg twice a day (BID) for 1 week, on gastric mucin production, the major component of mucus, in 20 asymptomatic volunteers and 20 patients with chronic constipation in basal conditions (primary outcome).

Specific Aim 4. To test the influence of Lubiprostone, 24 mcg twice a day (BID) for 1 week, on gastric mucin production, the major component of mucus, in 20 asymptomatic volunteers and 20 patients with chronic constipation during stimulation of gastric secretion with pentagastrin, mimicking the meal-stimulated conditions (primary outcome).

Specific Aim 5. To explore the impact of Lubiprostone, 24 mcg twice a day (BID) for 1 week, on viscoelasticity of gastric mucus in 20 asymptomatic volunteers and 20 patients with chronic constipation in basal conditions (secondary outcome).

Specific Aim 6. To address the impact of Lubiprostone, 24 mcg twice a day (BID) for 1 week, on viscoelasticity of gastric mucus in 20 asymptomatic volunteers and 20 patients with chronic constipation during stimulation of gastric secretion with pentagastrin, mimicking the meal-stimulated conditions (secondary outcome).

ELIGIBILITY:
Asymptomatic Volunteers:

Inclusion Criteria:

* 18-65 years of age
* Capable of and willing to give informed consent, and willing to comply with all study requirements

Exclusion Criteria:

* Pregnancy or lactation
* Subjects unwilling to practice adequate contraception throughout the screening period through 14 days after study termination
* Illegal use of illegal drugs
* Regular consumption of 2 or more drinks of alcohol per day
* Chronic non-steroidal anti- inflammatory drugs (NSAID) use
* Chronic use of H2 receptor antagonists or Proton Pump Inhibitors (PPIs) within 14 days prior to screening
* History of gastric of duodenal ulcer or chronic non-ulcer dyspepsia
* Positive Helicobacter pylori (H. pylori) serology

Patients with Chronic Constipation:

Inclusion Criteria:

* Age 18-65
* At least 6 months history of constipation. Constipation defined as: a. Less than three complete spontaneous bowel movements per week and one or more of the following: i) At least 25% of stools are very hard and/or hard stools ii) Sensation of incomplete evacuation following at least 25% of bowel movements iii) Straining on at least 25% of defecations The above criteria are only applicable to spontaneous bowel movements. Patients who have no spontaneous bowel movements (bowel movements are preceded by laxative intake) are considered constipated and are eligible for this study
* For patients >= years of age, normal colonic anatomy as documented by colonoscopy, double-contrast barium enema, or flexible sigmoidoscopy performed within the previous 5 years

Exclusion Criteria

* Pregnancy or lactation
* Subjects unwilling to practice adequate contraception throughout the period of screening through 14 days after study termination
* Use of laxatives 3 days immediately prior to randomization (except fiber or bulking agents)
* Use of any of the following drugs within 3 days prior to randomization a) Prokinetic agents (tegaserod, domperidone, cisapride, metoclopramide, erythromycin, b) Medications containing opiates c) Antispasmodic (e.g. atropine, hyoscyamine, scopolamine, glycopyrrolate)
* Use of illegal drugs
* Regular consumption of 2 drinks of alcohol per day
* Chronic NSAIDs use
* Chronic use of H2 receptor antagonist or PPIs within 14 days prior to screening
* History of gastric or duodenal ulcer, Inflammatory bowel disease (IBD), or chronic non-ulcer dyspepsia
* Diabetes mellitus (DM) type 1
* Parkinson's disease
* Existence of any medical condition that requires chronic therapy
* Positive H. pylori serology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Sarosiek, MD, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During an entire recruitment time all patients signed their consent forms and participate in the study protocol within the specially designated clinical research room at Texas Tech University Health Sciences Center(TTUHSC), El Paso.
Pre-assignment Details: Patients interested in our study were interviewed and examined 1 week before the 1st assigned after randomization medication was administered for one week of therapy.
  Subsequently, when patients finished their first week of medication, they had one week as of wash-out before the 2nd therapy in this cross-over design of our study protocol.
Groups:
- Chronic Constipation (CC)Subjects on Lubiprostone Then Placebo: Subjects with chronic constipation received 1 week of therapy with lubiprostone,then washed out for 1 week, then received 1 week of therapy with placebo.
  lubiprostone: 24mcg twice a day (BID)for 1 week; placebo pill: twice a day (BID) for 1 week
- Chronic Constipation (CC)Subjects on Placebo Then Lubiprostone: Subjects with chronic constipation received 1 week of therapy with placebo,then washed out for 1 week, then received 1 week of therapy with lubiprostone.
  placebo pill: twice a day (BID) for 1 week; lubiprostone: 24mcg twice a day (BID)for 1 week
- Controls on Lubiprostone Then Placebo: Control group received 1 week of therapy with lubiprostone, then washed out for 1 week, then received 1 week of therapy with placebo.
  lubiprostone: 24mcg twice a day (BID)for 1 week; placebo pill: twice a day (BID) for 1 week
- Controls on Placebo Then Lubiprostone: Control group received 1 week of therapy with placebo,then washed out for 1 week, then received 1 week of therapy with lubiprostone.
  placebo pill: twice a day (BID) for 1 week; lubiprostone: 24mcg twice a day (BID)for 1 week
Period: First Intervention
Arm/Group | Chronic Constipation (CC)Subjects on Lubiprostone Then Placebo | Chronic Constipation (CC)Subjects on Placebo Then Lubiprostone | Controls on Lubiprostone Then Placebo | Controls on Placebo Then Lubiprostone
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period for 1 Week
Arm/Group | Chronic Constipation (CC)Subjects on Lubiprostone Then Placebo | Chronic Constipation (CC)Subjects on Placebo Then Lubiprostone | Controls on Lubiprostone Then Placebo | Controls on Placebo Then Lubiprostone
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Chronic Constipation (CC)Subjects on Lubiprostone Then Placebo | Chronic Constipation (CC)Subjects on Placebo Then Lubiprostone | Controls on Lubiprostone Then Placebo | Controls on Placebo Then Lubiprostone
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Chronic Constipation(CC) Subjects on Lubiprostone Then Placebo: Subjects with chronic constipation (CC) received 1 week of therapy with lubiprostone, then washed out for 1 week, then received 1 week of therapy with placebo.
  lubiprostone: 24mcg twice a day (BID)for 1 week; placebo pill: twice a day (BID) for 1 week
- Chronic Constipation (CC)Subjects on Placebo Then Lubiprostone: Subjects with chronic constipation (CC)received 1 week of therapy with placebo,then washed out for 1 week, then received 1 week of therapy with lubiprostone.
  placebo pill: twice a day (BID) for 1 week; lubiprostone: 24mcg twice a day (BID)for 1 week
- Controls on Placebo Then Lubiprostone: Control group received 1 week of therapy with lubiprostone, then washed out for 1 week, then received 1 week of therapy with placebo.
  lubiprostone: 24mcg twice a day (BID)for 1 week; placebo pill: twice a day (BID) for 1 week
- Total: Total of all reporting groups
Arm/Group | Chronic Constipation(CC) Subjects on Lubiprostone Then Placebo | Chronic Constipation (CC)Subjects on Placebo Then Lubiprostone | Controls on Lubiprostone Then Placebo | Controls on Placebo Then Lubiprostone | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (16) | 37 (16) | 42 (18) | 42 (18) | 40 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 7 | 30
  Male | 2 | 3 | 2 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change of Mucus and Mucin Secretion in Patients With Chronic Constipation and in Controls.
Description: The rate of mucus and mucin secretion(mg/hr) will be measured in gastric juice aspirated in basal conditions and during stimulation with pentagastrin after 1 week of therapy with lubiprostone (Active Comparator) and compared with 1 week of placebo administration (Placebo Comparator).
Time Frame: Measured after 1 week of lubiprostone and 1 week of placebo with 1 week of washout period in between.
Population: Number of participants was calculated to provide statistical power of 0.80 for detection of significance.
Measure: Mean (Standard Error); unit: mg/hour
Groups:
- Lubiprostone 24 mcg BID; Placebo: Both controls and patients with chronic constipation received 1 week of therapy with lubiprostone (24 mcg twice a day)and 1 week of placebo (twice a day) in crossover design
Arm/Group | Lubiprostone 24 mcg BID | Placebo
Number analyzed (Participants) | 40 | 40
mg/hour
  Mucus Secretion in Chronic Constipation Subjects | 260 (29) | 133 (16)
  Mucus Secretion in Controls | 229 (33) | 161 (25)
  Mucin Secretion in Chronic Constipation Subjects | 99 (14) | 54 (7)
  Mucin Secretion in Controls | 100 (16) | 69 (14)

2. Secondary Outcome: Change in Viscoelasticity of Gastric Secretion in Controls and Patients With Chronic Constipation.
Description: The viscoelasticity of gastric mucus(centipoises) was measured in gastric juice aspirated in basal conditions and during stimulation with pentagastrin after 1 week of therapy with lubiprostone (Active Comparator) and compared with 1 week of placebo administration (Placebo Comparator).
Time Frame: Measured after 1 week of lubiprostone therapy and compared to 1 week of placebo with 1 week of washout in between.
Population: To provide 0.80 statistical power for detection of significance.
Measure: Mean (Standard Error); unit: Centipoises
Groups:
- Lubiprostone 24 mcg Bid: Both controls and patients with chronic constipation received lubiprostone 24 mcg twice daily for one week and placebo pills twice daily for one week in cross over design.
- Placebo: Both controls and patients with chronic constipation received lubiprostone 24mcg twice daily for one week and placebo pills twice daily for one week in cross over design.
Arm/Group | Lubiprostone 24 mcg Bid | Placebo
Number analyzed (Participants) | 40 | 40
Centipoises
  Basal viscosity in chronic constipation subjects | 21.61 (2.95) | 6.34 (1.01)
  Basal viscosity in controls | 12.78 (2.53) | 9.41 (1.74)
  Pentagastrin-Stimulated viscosity in CC | 14.96 (3.00) | 4.59 (1.20)
  Pentagastrin-Stimulated viscosity in Controls | 10.58 (2.20) | 7.84 (1.71)

ADVERSE EVENTS:
Groups:
- Chronic Constipation Subjects on Lubiprostone Then Placebo: Subjects with chronic constipation who received 1 week of therapy with lubiprostone, then washed out for 1 week, then received 1 week of therapy with placebo.
- Chronic Constipation Subjects on Placebo Then Lubiprostone: Subjects with chronic constipation who received 1 week of therapy with placebo, then washed out for 1 week, then received 1 week of therapy with lubiprostone.
- Controls on Lubiprostone Then Placebo: Control group who received 1 week of therapy with lubiprostone, then washed out for 1 week, then received 1 week of therapy with placebo.
- Controls on Placebo Then Lubiprostone: Control group who received 1 week of therapy with placebo, then washed out for 1 week, then received 1 week of therapy with lubiprostone.
Arm/Group | Chronic Constipation Subjects on Lubiprostone Then Placebo | Chronic Constipation Subjects on Placebo Then Lubiprostone | Controls on Lubiprostone Then Placebo | Controls on Placebo Then Lubiprostone
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No